CLINICAL TRIAL: NCT03573323
Title: A 24-Week Multicenter, Randomized, Blinded, Parallel-Group Study Comparing the Efficacy and Safety of Ixekizumab to Guselkumab in Patients With Moderate-to-Severe Plaque Psoriasis
Brief Title: A Study of Ixekizumab (LY2439821) Compared to Guselkumab in Participants With Moderate-to-Severe Plaque Psoriasis
Acronym: IXORA-R
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17119; I1F-MC-RHCR (Other: Eli Lilly and Company)
Record Dates: First submitted 2018-06-20; First posted 2018-06-29 (Actual); Results first posted 2020-07-28 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-02

CONDITIONS: Plaque Psoriasis
Keywords: biologic; biologic therapy
MeSH Terms: interventions — ixekizumab; guselkumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ixekizumab (Experimental): A starting dose of 160 milligram (mg) of ixekizumab was given as 2 subcutaneous (SC) injections at Week 0. During the Induction Period, ixekizumab 80 mg was given every 2 weeks (Q2W) at Weeks 2, 4, 6, 8, 10, and 12. During the Extension Period, ixekizumab 80 mg was given as 1 SC injection (Q4W) every 4 weeks at Weeks 16 and 20.
  The Post Treatment Follow Up Period was for safety monitoring following the last treatment period.
  Interventions: Drug: Ixekizumab
- Guselkumab (Experimental): During the Induction Period, guselkumab 100 mg was given as 1 SC injection at Weeks 0, 4 and 12. 1 placebo injection (to maintain the blind) was given at Weeks 0, 2, 6, 8, and 10. During the Extension Period, guselkumab 100 mg was given at Week 20. 1 placebo injection (to maintain the blind) was given at Week 16.
  The Post Treatment Follow Up Period was for safety monitoring following the last treatment period.
  Interventions: Drug: Guselkumab; Drug: Placebo

INTERVENTIONS:
Drug: Ixekizumab — Administered SC
  Other Names: LY2439821
  Arms: Ixekizumab
Drug: Guselkumab — Administered SC
  Arms: Guselkumab
Drug: Placebo — Administered SC
  Arms: Guselkumab

SUMMARY:
The purpose of this study is to compare the efficacy and safety of ixekizumab to guselkumab in participants with moderate-to-severe plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Have chronic plaque psoriasis based on a diagnosis for at least 6 months before baseline as determined by the investigator.
* Are a candidate for phototherapy and/or systemic therapy.
* Have both an Static Physician Global Assessment (sPGA) score of ≥3 and a Psoriasis Area and Severity Index (PASI) score ≥12 at screening and at baseline.
* Have ≥10% body surface area (BSA) involvement at screening and baseline.
* If a male, agree to use a reliable method of birth control during the study.
* If female, agree to use highly effective method of contraception.

Exclusion Criteria:

* Predominant pattern of pustular, erythrodermic, and/or guttate forms of psoriasis.
* Have a history of drug-induced psoriasis.
* Had a clinically significant flare of psoriasis during the 12 weeks before baseline.
* Use of tanning booths for at least 4 weeks before baseline.
* Concurrent or recent use of any biologic agent within the following periods prior to baseline: etanercept <28 days; infliximab, adalimumab, certolizumab pegol, or alefacept <60 days; golimumab <90 days; rituximab <12 months; secukinumab <5 months; or any other biologic agent (e.g., ustekinumab) <5 half lives.
* Have prior use of IL-23p19 antagonists (e.g., guselkumab, tildrakizumab, risankizumab), or have any condition or contraindication as addressed in the local labeling for guselkumab that would preclude the participant from participating in this protocol.
* Have previously completed or withdrawn from this study, participated in any other study with ixekizumab or guselkumab, have participated in any study investigating IL-23p19 antagonists, or have received treatment with ixekizumab.
* Have previously failed to respond to an IL-17 antagonist, per investigator assessment.
* Have had a live vaccination within 12 weeks of baseline.
* Have a known allergy or hypersensitivity to any biologic therapy.
* Have had any major surgery within 8 weeks of baseline.
* Have had a serious infection, have been hospitalized, or have received intravenous antibiotics for an infection within 12 weeks of baseline.
* Are women who are pregnant, or who are lactating (breast-feeding).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1027 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2020-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (124):
- United States (98):
  - Total Skin and Beauty Dermatology Center PC, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Alliance Dermatology and Mohs Center, Phoenix, Arizona
  - Perseverance Research Center, Scottsdale, Arizona
  - Johnson Dermatology, Fort Smith, Arkansas
  - Bakersfield Dermatology and Skin Cancer Medical Group, Bakersfield, California
  - Wallace Medical Group, Inc., Beverly Hills, California
  - California Dermatology and Clinical Research Institute, Encinitas, California
  - Tien Q. Nguyen, MD inc. DBA First OC Dermatology, Fountain Valley, California
  - Center for Dermatology Clinical Research, Inc., Fremont, California
  - Advanced Research Center, Los Alamitos, California
  - Axis Clinical Trials, Los Angeles, California
  - Dermatology Clinical Trials, Newport Beach, California
  - Quest Dermatology Research, Northridge, California
  - Northern California Research Corporation, Sacramento, California
  - Advanced Research Center, San Diego, California
  - Medical Center for Clinical Research, San Diego, California
  - University Clinical Trials, Inc., San Diego, California
  - Synergy Dermatology, San Francisco, California
  - Southern California Dermatology, Santa Ana, California
  - Mosaic Dermatology, Santa Monica, California
  - Clinical Science Institute, Santa Monica, California
  - Unison Clinical Trials, Sherman Oaks, California
  - Care Access Research-Walnut Creek, Walnut Creek, California
  - Dermatology Physicians of Connecticut, Shelton, Connecticut
  - Florida Academic Dermatology Centers, Coral Gables, Florida
  - Olympian Clinical Research, Largo, Florida
  - Suncoast Research Group, LLC, Miami, Florida
  - Miami Dermatology & Laser Research, Miami, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - Renstar Medical Research, Ocala, Florida
  - Sensible Healthcare, Ocoee, Florida
  - Park Avenue Dermatology, Orange Park, Florida
  - International Clinical Research, Sanford, Florida
  - MOORE Clinical Research, Tampa, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Olympian Clinical Research, Tampa, Florida
  - Atlanta Dermatology, Vein Research Center, PC, Alpharetta, Georgia
  - Skin Care Physicians of Georgia, Macon, Georgia
  - Arlington Dermatology, Rolling Meadows, Illinois
  - Dermatology Institute of Dupage Medical Group, Wheaton, Illinois
  - Qualmedica Research LLC, Evansville, Indiana
  - Dawes Fretzin Clinical Research, Indianapolis, Indiana
  - Dermatology Specialists Research Indiana, New Albany, Indiana
  - The Indiana Clinical Trials Center, PC, Plainfield, Indiana
  - The South Bend Clinic, South Bend, Indiana
  - Integrated Clinical Trial Services, Inc., West Des Moines, Iowa
  - Kansas City Dermatology, PA, Overland Park, Kansas
  - Dermatology Specialist, Louisville, Kentucky
  - Owensboro Dermatology Associates, Owensboro, Kentucky
  - Lawrence J Green, M.D, LLC, Rockville, Maryland
  - ActivMed Practices & Research, Inc, Beverly, Massachusetts
  - Fivenson Dermatology, Ann Arbor, Michigan
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - Clarkston Skin Research, Clarkston, Michigan
  - Henry Ford Medical Center- New Center One, Detroit, Michigan
  - St Joseph Dermatology and Vein Clinic, Saint Joseph, Michigan
  - Central Dermatology PC, St Louis, Missouri
  - Impact Clinical Trials, Las Vegas, Nevada
  - ActivMed Practices & Research, Inc, Portsmouth, New Hampshire
  - Psoriasis Treatment Center of Central New Jersey, East Windsor, New Jersey
  - Forest Hills Dermatology Group, Forest Hills, New York
  - Sadick Research Group, New York, New York
  - Piedmont Plastic Surgery and Dermatology, Charlotte, North Carolina
  - Dermatology Consulting Services, High Point, North Carolina
  - PMG Research of Rocky Mount, LLC, Rocky Mount, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Bexley Dermatology Research, Bexley, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Wright State Univ School of Medicine, Fairborn, Ohio
  - Ohio State Univ College Of Medicine, Gahanna, Ohio
  - Dermatologists of Southwest Ohio, Inc., Mason, Ohio
  - Oregon Medical Research Center, Portland, Oregon
  - Dermatology and Skin Surgery Center, Exton, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Yardley Dermatology, Yardley, Pennsylvania
  - Clinical Partners LLC, Johnston, Rhode Island
  - Clinical Research Center of the Carolinas, Charleston, South Carolina
  - International Clinical Research, Murfreesboro, Tennessee
  - Arlington Research Center, Inc, Arlington, Texas
  - Austin Institute for Clinical Research, Inc., Austin, Texas
  - Bellaire Dermatology, Bellaire, Texas
  - Dermatology Treatment and Research Center, Dallas, Texas
  - Modern Research Associates PLLC, Dallas, Texas
  - Center for Clinical Studies, Houston, Texas
  - Suzanne Bruce and Associates, PA, Houston, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
  - Stephen L Miller, MD, PA, San Antonio, Texas
  - University of Utah MidValley Dematology, Murray, Utah
  - Virginia Clinical Research, Norfolk, Virginia
  - Virginia Dermatology & Skin Cancer Center, Norfolk, Virginia
  - Eastern Virginia Medical School, Norfolk, Virginia
  - National Clinical Research - Richmond, Richmond, Virginia
  - Dermatology Associates, Seattle, Washington
  - West Virginia Research Institute, Morgantown, West Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (20):
  - Dermatology Research Institute Inc., Calgary, Alberta
  - Kirk Barber Research, Calgary, Alberta
  - Stratica Medical, Edmonton, Alberta
  - Dr. Chih-ho Hong Medical Inc., Surrey, British Columbia
  - Enverus Medical Research, Surrey, British Columbia
  - Wiseman Dermatology Research Inc., Winnipeg, Manitoba
  - Karma Clinical Trials Inc, St. John's, Newfoundland and Labrador
  - Eastern Canada Cutaneous Research Assoicates Ltd, Halifax, Nova Scotia
  - Dermatrials Research Inc., Hamilton, Ontario
  - Mediprobe Research Inc, London, Ontario
  - The Guenther Dermatology Research Centre, London, Ontario
  - Lynderm Research Inc, Markham, Ontario
  - DermEdge Research Inc, Mississauga, Ontario
  - North Bay Dermatology Centre, North Bay, Ontario
  - SKiN Centre for Dermatology, Peterborough, Ontario
  - The Centre for Dermatology, Richmond Hill, Ontario
  - K. Papp Clinical Research Inc, Waterloo, Ontario
  - Dr Isabelle Delorme Inc., Drummondville, Quebec
  - Innovaderm Research Inc, Montreal, Quebec
  - Q&T Research Sherbrooke Inc, Sherbrooke, Quebec
- Puerto Rico (6):
  - Centro Reumatologico de Caguas, Caguas, PR
  - Office of Dr. Samuel Sanchez PSC, Caguas, PR
  - Ponce School of Medicine CAIMED Center, Ponce, PR
  - GCM Medical Group PSC, San Juan, PR
  - Mindful Medical Research, San Juan, PR
  - Santa Cruz Behavioral PSC, Bayamón

IPD SHARING:
Plan to Share IPD: Yes
Lilly provides access to the individual patient data from studies on approved medicines and indications as defined by the sponsor specific information on ClinicalStudyDataRequest.com This access is provided in a timely fashion after the primary publication is accepted. Researchers need to have an approved research proposal submitted through ClinicalStudyDataRequest.com. Access to the data will be provided in a secure data sharing environment after signing a data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org

REFERENCES:
- [Derived] Armstrong A, Gonzalez-Cantero A, Khattri S, Muzy G, Malatestinic WN, Lampropoulou A, Feely M, See SK, Mert C, Blauvelt A. Comparing Achievement of National Psoriasis Foundation Treatment Targets among Patients with Plaque Psoriasis Treated with Ixekizumab versus Other Biologics in Clinical and Real-World Studies. Dermatol Ther (Heidelb). 2024 Apr;14(4):933-952. doi: 10.1007/s13555-024-01136-w. Epub 2024 Mar 23. PMID 38521874
- [Derived] Gooderham M, Vender R, Crowley J, Hong HC, Feely M, Garrelts A, See K, Konicek B, Green L. Speed and Cumulative Responses According to Body Regions in Patients with Moderate-to-Severe Plaque Psoriasis Treated with Ixekizumab (Interleukin-17A Antagonist) versus Guselkumab (Interleukin-23p19 Inhibitor). Dermatol Ther (Heidelb). 2024 Feb;14(2):441-451. doi: 10.1007/s13555-023-01075-y. Epub 2024 Feb 9. PMID 38332436
- [Derived] Elewski BE, Blauvelt A, Gallo G, Wolf E, McKean-Matthews M, Burge R, Merola JF, Gottlieb AB, Guenther LC. Simultaneous Nail and Skin Clearance in Ixekizumab Head-to-Head Trials for Moderate-to-Severe Psoriasis and Psoriatic Arthritis. Dermatol Ther (Heidelb). 2022 Apr;12(4):911-920. doi: 10.1007/s13555-022-00704-2. Epub 2022 Mar 13. PMID 35279805
- [Derived] Blauvelt A, Leonardi C, Elewski B, Crowley JJ, Guenther LC, Gooderham M, Langley RG, Vender R, Pinter A, Griffiths CEM, Tada Y, Elmaraghy H, Lima RG, Gallo G, Renda L, Burge R, Park SY, Zhu B, Papp K; IXORA-R Study Group. A head-to-head comparison of ixekizumab vs. guselkumab in patients with moderate-to-severe plaque psoriasis: 24-week efficacy and safety results from a randomized, double-blinded trial. Br J Dermatol. 2021 Jun;184(6):1047-1058. doi: 10.1111/bjd.19509. Epub 2020 Oct 25. PMID 32880909

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consists of a combined blinded treatment (trt) period with a 24-week duration followed by a post treatment follow-up (PTFU) period with a minimum of a 12-week duration. The Induction Dosing Period (12 Weeks) and Extension Period (12 Weeks) were combined for analysis and referred to as the blinded treatment periods.
Period: Blinded Treatment Period (Weeks 0-24)
Arm/Group | Ixekizumab | Guselkumab
Started | 520 | 507
Received at Least One Dose of Study Drug | 519 | 506
Completed | 465 | 459
Not Completed | 55 | 48
Not completed — Screen Failure | 1 | 1
Not completed — Adverse Event | 15 | 8
Not completed — Protocol Violation | 3 | 8
Not completed — Withdrawal by Subject | 17 | 9
Not completed — Lack of Efficacy | 2 | 3
Not completed — Pregnancy | 1 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 14 | 13
Not completed — Sponsor Decision | 0 | 1
Not completed — Alkaline Phosphatase (ALP) level reached | 0 | 1
Not completed — Noncompliant to protocol procedures | 1 | 2
Period: Post-Treatment Follow Up (Weeks 25-36)
Arm/Group | Ixekizumab | Guselkumab
Started | 465 | 456 (Excludes participants who completed treatment and did not enter the PTFU.)
Completed | 406 | 399
Not Completed | 59 | 57
Not completed — Withdrawal by Subject | 22 | 12
Not completed — Lack of Efficacy | 8 | 19
Not completed — Physician Decision | 4 | 3
Not completed — Did not wish to return to study | 3 | 2
Not completed — Discontinued Trt and Completed Follow Up | 14 | 8
Not completed — Not Compliant to Protocol Procedures | 8 | 11
Not completed — Sponsor Decision | 0 | 1
Not completed — Repeat Infections | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ixekizumab | Guselkumab | Total
Number analyzed (Participants) | 520 | 507 | 1027
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: All randomized participants who received at least one dose of study drug and had baseline Age data.
  years
    number analyzed (Participants) | 519 | 506 | 1025
    (all) | 49.0 (13.90) | 49.0 (14.88) | 49.0 (14.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 182 | 193 | 375
  Male | 338 | 314 | 652
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 127 | 120 | 247
  Not Hispanic or Latino | 383 | 379 | 762
  Unknown or Not Reported | 10 | 8 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 6 | 13
  Asian | 31 | 35 | 66
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
  Black or African American | 38 | 29 | 67
  White | 439 | 431 | 870
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 103 | 106 | 209
  United States | 417 | 401 | 818

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving 100% Improvement From Baseline in Psoriasis Area and Severity Index (PASI 100)
Description: The PASI combines assessments of the extent of body-surface involvement in 4 anatomical regions (head, trunk, arms, and legs) and the severity of desquamation (scaling), erythema, and plaque induration/infiltration (thickness) in each region, yielding an overall score of 0 for no psoriasis to 72 for the most severe disease. Participants achieving PASI 100 were defined as having an improvement of at least 100% in the PASI scores compared to baseline.
Time Frame: Week 12
Population: All randomized participants. Participants who did not meet clinical response criteria or have missing data at Week 12 were considered as non-responders for the Non-Responder Imputation (NRI) analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Ixekizumab: A starting dose of 160 milligram (mg) of ixekizumab was given as 2 subcutaneous (SC) injections at Week 0. During the Induction Period, ixekizumab 80 mg was given every 2 weeks (Q2W) at Weeks 2, 4, 6, 8, 10, and 12. During the Extension Period, ixekizumab 80 mg was given as 1 SC injection (Q4W) every 4 weeks at Weeks 16 and 20. The Post Treatment Follow Up Period was for safety monitoring following the last treatment period and study visit.
- Guselkumab: During the Induction Period, guselkumab 100 mg was given as 1 SC injection at Weeks 0, 4 and 12. 1 placebo injection (to maintain the blind) was given at Weeks 0, 2, 6, 8, and 10. During the Extension Period, guselkumab 100 mg was given at Week 20. 1 placebo injection (to maintain the blind) was given at Week 16. The Post Treatment Follow Up Period was for safety monitoring following the last treatment period and study visit.
Arm/Group | Ixekizumab | Guselkumab
Number analyzed (Participants) | 520 | 507
percentage of participants | 41.3 [37.1 to 45.6] | 24.9 [21.1 to 28.6]
Statistical Analysis 1: Comparison: Ixekizumab vs Guselkumab; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel

2. Secondary Outcome: Percentage of Participants Achieving PASI 75
Description: The PASI combines assessments of the extent of body-surface involvement in 4 anatomical regions (head, trunk, arms, and legs) and the severity of desquamation (scaling), erythema, and plaque induration/infiltration (thickness) in each region, yielding an overall score of 0 for no psoriasis to 72 for the most severe disease. Participants achieving PASI 75 were defined as having an improvement of at least 75% in the PASI scores compared to baseline.
Time Frame: Week 2
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ixekizumab | Guselkumab
Number analyzed (Participants) | 520 | 507
percentage of participants | 22.9 [19.3 to 26.5] | 5.1 [3.2 to 7.0]
Statistical Analysis 1: Comparison: Ixekizumab vs Guselkumab; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel

3. Secondary Outcome: Percentage of Participants Achieving PASI 90
Description: The PASI combines assessments of the extent of body-surface involvement in 4 anatomical regions (head, trunk, arms, and legs) and the severity of desquamation (scaling), erythema, and plaque induration/infiltration (thickness) in each region, yielding an overall score of 0 for no psoriasis to 72 for the most severe disease. Participants achieving PASI 90 were defined as having an improvement of at least 90% in the PASI scores compared to baseline.
Time Frame: Week 4
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ixekizumab | Guselkumab
Number analyzed (Participants) | 520 | 507
percentage of participants | 21.0 [17.5 to 24.5] | 7.9 [5.5 to 10.2]
Statistical Analysis 1: Comparison: Ixekizumab vs Guselkumab; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel

4. Secondary Outcome: Percentage of Participants Achieving PASI 100
Description: as for outcome 1
Time Frame: Week 4
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ixekizumab | Guselkumab
Number analyzed (Participants) | 520 | 507
percentage of participants | 6.7 [4.6 to 8.9] | 1.4 [0.4 to 2.4]
Statistical Analysis 1: Comparison: Ixekizumab vs Guselkumab; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel

5. Secondary Outcome: Percentage of Participants Achieving PASI 90
Description: as for outcome 3
Time Frame: Week 8
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ixekizumab | Guselkumab
Number analyzed (Participants) | 520 | 507
percentage of participants | 58.5 [54.2 to 62.7] | 35.9 [31.7 to 40.1]
Statistical Analysis 1: Comparison: Ixekizumab vs Guselkumab; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel

6. Secondary Outcome: Percentage of Participants Achieving Static Physician Global Assessment (sPGA) (0)
Description: The sPGA is a physician's determination of the participant's psoriasis lesions overall at a given time point categorized by descriptions for induration, erythema, and scaling. For the analysis of responses, the participant's psoriasis is assessed as clear (0), minimal (1), mild (2), moderate (3), severe (4), or very severe (5). An sPGA (0) response was defined as a post-baseline sPGA score of 0.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ixekizumab | Guselkumab
Number analyzed (Participants) | 520 | 507
percentage of participants | 41.9 [37.7 to 46.2] | 25.2 [21.5 to 29.0]
Statistical Analysis 1: Comparison: Ixekizumab vs Guselkumab; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel

7. Secondary Outcome: Percentage of Participants Achieving PASI 50
Description: The PASI combines assessments of the extent of body-surface involvement in 4 anatomical regions (head, trunk, arms, and legs) and the severity of desquamation (scaling), erythema, and plaque induration/infiltration (thickness) in each region, yielding an overall score of 0 for no psoriasis to 72 for the most severe disease. Participants achieving PASI 50 were defined as having an improvement of at least 50% in the PASI scores compared to baseline.
Time Frame: Week 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ixekizumab | Guselkumab
Number analyzed (Participants) | 520 | 507
percentage of participants | 27.5 [23.7 to 31.3] | 9.3 [6.7 to 11.8]
Statistical Analysis 1: Comparison: Ixekizumab vs Guselkumab; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel

8. Secondary Outcome: Percentage of Participants Achieving PASI 100
Description: as for outcome 1
Time Frame: Week 8
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ixekizumab | Guselkumab
Number analyzed (Participants) | 520 | 507
percentage of participants | 29.6 [25.7 to 33.5] | 13.6 [10.6 to 16.6]
Statistical Analysis 1: Comparison: Ixekizumab vs Guselkumab; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel

9. Secondary Outcome: Percentage of Participants Achieving PASI 100
Description: as for outcome 1
Time Frame: Week 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ixekizumab | Guselkumab
Number analyzed (Participants) | 520 | 507
percentage of participants | 50.0 [45.7 to 54.3] | 52.3 [47.9 to 56.6]
Statistical Analysis 1: Comparison: Ixekizumab vs Guselkumab; Test type: Superiority; p = 0.414, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: Up to 48 Weeks
Description: All randomized participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Groups:
- Ixekizumab Post-Treatment Follow Up: Participants who received ixekizumab in the blinded treatment periods entered the post treatment follow up period.
- Guselkumab Post-Treatment Follow Up: Participants who received guselkumab in the blinded treatment periods entered the post treatment follow up period.
Arm/Group | Ixekizumab | Guselkumab | Ixekizumab Post-Treatment Follow Up | Guselkumab Post-Treatment Follow Up
All-Cause Mortality (participants affected / at risk) | 0/519 | 0/506 | 0/465 | 0/456
Serious Adverse Events (participants affected / at risk) | 18/519 | 16/506 | 4/465 | 4/456
Other Adverse Events (participants affected / at risk) | 113/519 | 73/506 | 11/465 | 9/456
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Ixekizumab (N=519) | Guselkumab (N=506) | Ixekizumab Post-Treatment Follow Up (N=465) | Guselkumab Post-Treatment Follow Up (N=456)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Salivary gland calculus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Complicated appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endometrial cancer stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/182 (0) | 1/193 (1) | 0/164 (0) | 0/170 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhabdomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myxoedema coma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0/337 (0) | 0/313 (0) | 0/301 (0) | 1/286 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertensive urgency (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ixekizumab (N=519) | Guselkumab (N=506) | Ixekizumab Post-Treatment Follow Up (N=465) | Guselkumab Post-Treatment Follow Up (N=456)
Injection site reaction (General disorders) | 49 (80) | 6 (9) | 0 (0) | 1 (2)
Nasopharyngitis (Infections and infestations) | 34 (41) | 27 (29) | 5 (5) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 40 (44) | 41 (50) | 6 (6) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-12-07): https://cdn.clinicaltrials.gov/large-docs/23/NCT03573323/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-31): https://cdn.clinicaltrials.gov/large-docs/23/NCT03573323/SAP_001.pdf